CLINICAL TRIAL: NCT00590382
Title: Emergency/Compassionate Use - Muscular VSD Occluder
Status: Approved for marketing | Type: Expanded Access
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: AGA-005 - E/C; G990289
Record Dates: First submitted 2007-12-20; First posted 2008-01-10 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Muscular; Ventricular; Septal; Defects; VSD

INTERVENTIONS:
Device: AMPLATZER Muscular VSD Occluder — AMPLATZER Muscular VSD Occluder

SUMMARY:
Expanded access to the AMPLATZER Muscular VSD Occluder

ELIGIBILITY:
Inclusion Criteria:

* Emergency/compassionate use for patients not meeting the inclusion criteria for the AMPLATZER Muscular VSD clinical trial

Sex: All
Age Groups: Child, Adult, Older Adult